CLINICAL TRIAL: NCT05935046
Title: Effects of Hormonal STatus on Energy Expenditure and Feeding behAvior in woMen
Brief Title: Effects of Hormonal STatus on Energy Expenditure and Feeding behAvior in woMen(ESTEAM)
Acronym: ESTEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2022 DUCLOS 2; 2022-A02464-39 (Other: ANSM)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Energy Expenditure, Appetite, Energy Intake, Food Reward Menopause Transition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Premenopausal Status (Experimental)
  Interventions: Behavioral: Walk test and meal test
- Peri Menopausal status (Experimental)
  Interventions: Behavioral: Walk test and meal test
- Menopausal status (Experimental)
  Interventions: Behavioral: Walk test and meal test

INTERVENTIONS:
Behavioral: Walk test and meal test — The subjects will perform a treadmill walking test at increasing speed from 2 to 6km.h-1 in 5min increments.
  During the second experimental visit, subjects will be required to consume a test meal containing 590kcal (12% protein, 35% fat, 53% carbohydrate) (Duhita et al 2017).
  The composition of the test meal will be developed based on the food preferences and habits questionnaires completed during the inclusion visit. Foods indicated as "preferred" by participants will not be offered during these sessions to avoid any influence of their palatable nature on participants' consumption.

SUMMARY:
The health of women throughout their lives and especially during aging is a subject at the heart of current health issues. Indeed, hormonal variations during a woman's life condition her reproductive life, but also her cardiometabolic health (insulin sensitivity, lipid and inflammatory profile), musculoskeletal health and the maintenance of her mobility. The changes in body composition that occur with age, but also according to hormonal status (Isacco et al. 2021), as well as the metabolic impact of menopause are mechanisms favoring weight gain and more specifically fat mass (Leeners et al 2017). The decrease in estrogen levels during the transition to menopause seems to be the main factor explaining the increase in adiposity, especially visceral, and a decrease in muscle capital. Indeed, estrogens participate in the structural remodeling of muscle tissue as well as in maintaining its oxidative potential (Sutham et al 2018). However, the mechanisms promoting changes in body composition during the transition to menopause remain poorly understood. Better characterizing the energy profile (energy expenditure) and the food profile with regard to body composition in non- and postmenopausal women would make it possible to better target the recommendations for the primary prevention of cardiometabolic alterations linked to ovarian aging.

ELIGIBILITY:
Inclusion Criteria:

* Adult female volunteer
* Body mass index > 18.5 kg/m2 and ≤35 kg/m2
* Able to provide informed consent to participate in research
* Subject to a Social Security scheme.
* Pre-menopausal woman with or without oral contraception and having regular menstrual cycles (21-35 days) or
* Perimenopausal woman: presence of irregularity in the menstrual cycles (>7 days) and/or amenorrhea ≥2 and 12 months or
* Postmenopausal woman: amenorrhea (absence of menstruation) for at least one year and for a maximum of 10 years, and menopause having appeared after 40 years.

Exclusion Criteria:

* Chronic illness or a long-term condition, being under medical treatment
* Pregnant or breastfeeding women.
* Women on contraceptives other than oral contraceptives
* Postmenopausal women undergoing hormonal treatment for menopause
* Cardiorespiratory and/or osteo-articular disorders limiting their ability to perform the walk test
* Type 1 diabetes or type 2 diabetes treated with medication
* Progressive cardiovascular or neoplastic disease.
* Major infection in the 3 months preceding inclusion.
* Known neuromuscular pathology: myopathy, myasthenia, rhabdomyolysis, paraplegia, hemiplegia,
* Chronic or acute inflammatory disease in the 3 months preceding inclusion
* Treatment with beta-blocker
* Diagnosis or treatment for schizophrenia, bipolar disorder, major depression
* Discontinuation of treatment for less than 3 months prior to inclusion, with corticosteroids, immunosuppressant, anabolic, growth hormone.
* Eating behavior disorders
* Amenorrhea linked to a pathology or its treatment (pituitary tumour, radiotherapy, chemotherapy, oophorectomy, etc.)
* Unstable psychiatric state
* Significant alcohol consumption (> 2 to 3 drinks per day depending on gender) or the presence of drug addiction.
* Inability to walk for 30 minutes at a time
* Subject in a period of exclusion from another study or having received more than €4,500 in the year following their participation in clinical studies.
* Deprivation of liberty by judicial or administrative decision (guardianship, curatorship or safeguard of justice).
* Refusal to sign the written consent to participate.
* Participation in another study in the previous 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Resting energy expenditure and EE during the walk test will be assessed during the first experimental day. Thermic effect of food will be investigated during the second experimental day.
  Resting energy expenditure will be calculated, on an empty stomach, for 30 minutes using the indirect calorimetry method.
  Energy expenditure will be assessed during walking exercise by portable indirect calorimetry (MetaMax, Inc.) through the measurement of gas exchange. Indirect calorimetry is one of the classic methods of measuring energy expenditure during exercise.
  After the test meal, energy expenditure will be evaluated in the postprandial period by indirect calorimetry for 180 min (MétaMax, Inc.). During the measurement, the subject will be seated comfortably in an armchair and will be offered the opportunity to view a calm film/documentary throughout the measurement in order to limit boredom.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No